CLINICAL TRIAL: NCT05362916
Title: Influence of a 3-month Letermovir Treatment on Gut Inflammation in ART-treated HIV-infected Persons in an Open Labelled Controlled Randomized Study
Brief Title: Letermovir in ART-treated HIV-infected Persons
Acronym: Letermovir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean-Pierre Routy (Other)
Responsible Party: Sponsor-Investigator, Jean-Pierre Routy, Clinical Director of the Chronic Viral Illness Service Division of Hematology and Chronic Viral Illness Service Louis Lowenstein Chair in Hematology & Oncology Professor of Medicine, McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-37-2022-8295
Record Dates: First submitted 2022-04-22; First posted 2022-05-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: People Living With HIV
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Intervention Model Description: Multi-centre, open-label, randomized, controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letermovir (Experimental): 40 patients with CMV infection will be treated with Letermovir
  Interventions: Drug: Letermovir
- Controls (No Intervention): 20 patients with CMV infection will not be given Letermovir

INTERVENTIONS:
Drug: Letermovir — Participants in the treatment arm will take either 1 tablet of 480mg PO once daily or 2 tablets of 240mg PO once daily.
  Other Names: PREVYMIS
  Arms: Letermovir

SUMMARY:
This is a multi-centre, open-label, randomized, controlled clinical trial to assess the influence of letermovir on gut translocation marker LPS in blood in ART-treated cytomegalovirus (CMV)-seropositive adult people living with HIV (PLWH). The study will explore the influence of letermovir treatment on gut damage, with no intention for label change. Participants (n=60) should have a cluster of differentiation 4 cells (CD4) count greater than 400 cells/µl and a negative viral load. Forty (40) participants will be randomized to receive letermovir (PREVYMIS® 480 mg or 2x240mg orally) in addition to their usual ART, and 20 participants will receive standard of care alone (ART only) for 14 weeks. Study visits will include screening, 2 baselines, followed by follow-up visits at 2 and 4 weeks and at 14 weeks after starting treatment and 12 weeks after end of letermovir treatment to assess a carry-over effect.

In an optional sub-study, colonoscopies and colon biopsies will be performed before and after letermovir treatment or standard of care alone to assess gut mucosa inflammation.

DETAILED DESCRIPTION:
INTRODUCTION, BACKGROUND, AND STUDY RATIONALE

Cytomegalovirus (CMV) seropositivity is frequent in the general population and even more so in persons living with HIV (PLWH). In the general population, high anti-CMV immunoglobulins G (IgG)-titer has been associated with earlier mortality, cluster of differentiation 8 (CD8) T-cell expansion, low CD4/CD8 ratio and increased cluster of differentiation cells (CD57) senescence marker expression on T cells. Such elevated IgG titer may be linked to transient CMV replication. The investigators have shown that gut permeability is correlated with anti-CMV IgG titers in PLWH on antiretroviral therapy (ART). Increased gut permeability is associated with microbial translocation and systemic inflammation, and correlates with frequency of non-infectious/non-AIDS comorbidities such as cardiovascular diseases, neurocognitive disorders and cancer. Moreover, gut permeability has been linked with reduced response to commercialized vaccines . The investigators recently demonstrated that, in HIV elite controllers, a rare subgroup of PLWH who can control HIV replication in absence of ART, CMV coinfection and anti-CMV IgG levels were associated with CD4 count decay. As HIV replication is well controlled with ART, our findings suggest that CMV co-infection is a driving factor behind increased gut permeability and inflammation in PLWH, contributing to immune exhaustion and senescence.

Hunt et al. have shown that administration of valganciclovir, an anti-CMV medication, in ART-treated PLWH for 4 weeks was associated with a decrease in immune activation markers compared to the control group. However, long-term use of valganciclovir is not convenient due to its toxicity and its activity is not specific to CMV. Furthermore, its influence on gut permeability has not been assessed.

A novel anti-CMV agent with an excellent safety profile, letermovir, was approved in 2017 for anti-CMV prophylaxis in allogeneic hematopoietic cell transplant recipients. In these patients, a drastic reduction of both low-grade replication and CMV infections, combined with an improved immune reconstitution after the graft was reported. In vitro, in intestinal tissues reconstituted from primary cells, letermovir anti-CMV treatment could prevent CMV-induced epithelial disruption.

Potential Risks and Benefits to Human Participants

Potential Risks Associated with letermovir

For this study, participants will be receiving two tablets of 240mg or one tablet of 480mg of PREVYMIS® daily, for 14 weeks in total. This corresponds to the dose recommended for anti-CMV prophylaxis in hematopoietic cell transplant recipients. In this latter population, which is the only one for which PREVYMIS® has been approved in Canada, most frequent side effects are nausea/vomiting and peripheral edema. Cardiac events constitute 13% of all adverse effects, including atrial fibrillation in 3.5, as such an ECG will be performed during the screening visit and participants with any type of known arrythmia will be excluded. In case of cardiac symptoms during follow-up, another ECG will be performed and participants with arrythmia will be withdrawn from the study and referred to a cardiologist. In practice, those side effects are unfrequent, as illustrated in the pivotal clinical trial of letermovir in which frequency and severity of adverse events were not statistically increased in the letermovir group compared to placebo group.

Finally, based on the Canadian PREVYMIS® monograph, drug-on-drug interactions are possible and the concomitant administration of following medications will constitute exclusion criteria: pimozide, ergotamine, lovastatin, rosuvastatin, simvastatin or bosentan when co-administered with cyclosporine. For patients not using cyclosporine, dose of statins will be reduced by 50% for the duration of the letermovir or placebo treatment. Due to the long-term effect of statins, such a short-period of dose reduction is not expected to increase cardiovascular risk to participants. Regarding HIV medication, exclusionary agents include darunavir, efavirenz, etravirine and nevirapine. Those drugs constitute parts of ART regimens and participants who receive them will need to be excluded. However, this should not significantly impact recruitment as these drugs are only rarely prescribed in HIV clinics in Quebec.

Exclusionary agents have been discussed and accepted by the Merck Investigator Studies Program Safety Committee of Merck.

Potential risks to blood draws

The risks of drawing blood from a vein include: discomfort at the blood draw site (often momentary); possible bruising, redness, swelling, and/or bleeding at the site (will be managed by putting pressure on site of draw); feeling of lightheadedness when blood is drawn (will be managed by ensuring participants remains seated until dizziness abates); and rarely an infection at the site where the blood was drawn (cleaning of the site prior to blood draw should prevent this from happening, and treatment in case of infection will be provided).

Potential risks and/or discomforts to colon mucosal biopsies

Participants from McGill University Health Centre (MUHC) will be invited to participate in an optional sub-study to collect colon mucosal biopsy. They will be asked to sign a separate consent form if they wish to take part in the sub-study.

The day before this procedure, the consenting participant will be required to take measures to clear his/her bowels for the examination by drinking a picosulfate based solution and magnesium citrate as enunciated in the colonoscopy information preparation sheet (Appendix 5).

The Information sheet addendum will be given to each participant referring side effects, risks, contraindications and the medication interactions for the two magnesium-based products used to clean their bowels.

During the colon mucosal biopsy procedure, the participant may feel pressure in the rectum similar to the sensation felt with the urge to have a bowel movement. The participant may also feel a small amount of abdominal cramping. The most serious risk of the procedure is perforation, i.e. poking a hole in the lining of the intestine; this risk is extremely uncommon, occurring once out of every 10,000 procedures. Some bleeding will likely occur at the place where the biopsies are done. Light to moderate sedation using midazolam and fentanyl could be used during the procedure, in the absence of any contraindication. This sedation procedure is very safe, rare side effects include temporary memory loss, blood pressure drop or vomiting. If the participant experiences severe discomfort despite sedation during the colon mucosal biopsies, the procedure will be stopped immediately; he/she will be seen by a physician and the research nurse will monitor him/her until he/she is ready to go home.

1.3.4 Benefits to Participating in This Study

The effects of CMV latent infection has been widely reported and include persisting inflammation, gut leakage, decreased response to vaccines and to pathogens. As such, a potential beneficial effect of letermovir on those parameters is expected, which is particularly meaningful in the light of the current COVID-19 pandemic. Altogether, findings from this study may clarify the influence of CMV on health, and help to improve treatments for PLWH. The study's results will be published and all participants will be given access to the study findings.

Study Rationale

Latent CMV infection and occasional replication has been linked with poorer outcome in PLWH. Our hypothesis is that inhibiting CMV replication with a safe anti-CMV agent as letermovir will prevent gut damage and favor gut epithelium repair, decreasing microbial translocation and lower non-AIDS comorbidity risks in ART-treated PLWH.

Based on our experience, and recent trials such at the single arm Clinical Trials Network (CTN) PT27 Lilac study, the investigators propose a randomized controlled trial with a control arm receiving standard of care (ART only) to ensure the specificity of any changes the investigators could observe with letermovir (long term ART treatment could influence inflammation markers). Such a design is optimal for the development of future larger studies, in the case where results would show a clinical interest.

STUDY OBJECTIVES AND DESIGN

Overall Study Design

This is a multi-centre, open-label, randomized, controlled clinical trial to assess the influence of letermovir on gut translocation marker LPS in blood in ART-treated CMV-seropositive adult PLWH. The study will explore the influence of letermovir treatment on gut damage, with no intention for label change. Participants (n=60) should have a CD4 count greater than 400 cells/µl and a negative viral load. Forty (40) participants will be randomized to receive letermovir (PREVYMIS® 480 mg or 2x240mg orally) in addition to their usual ART, and 20 participants will receive standard of care alone (ART only) for 14 weeks. Study visits will include screening, 2 baselines, followed by follow-up visits at 2 and 4 weeks and at 14 weeks after starting treatment and 12 weeks after end of letermovir treatment to assess a carry-over effect.

In an optional sub-study, colonoscopies and colon biopsies will be performed before and after letermovir treatment or standard of care alone to assess gut mucosa inflammation.

Primary Objective(s)

To assess the influence of CMV replication inhibition with letermovir on gut translocation markers (LPS) in blood of PLWH.

Secondary Objective(s)

To assess the influence of CMV replication inhibition with letermovir on:

Gut permeability markers in blood of PLWH (REG3α and I-FABP). Inflammation markers (IL-6, sCD14, hsCRP, d-dimers) in blood of PLWH. Anti-CMV immune response (anti-CMV IgG titers and specific T-cell response) and CMV DNA detection in plasma and Peripheral Blood Mononuclear Cells (PBMC).

In a sub-study, inflammation in colon biopsies obtained by coloscopy and in CMV DNA detection in gut mucosa

Exploratory Objectives(s)

To assess the influence of CMV replication inhibition with letermovir on:

HIV reservoir size in blood and mucosal samples. Microbiota composition.

Sub-studies

In an optional sub-study, colonoscopies and colon biopsies will be performed before and after letermovir treatment or standard of care alone to assess gut mucosa inflammation.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible for the study if they meet the following criteria:

1. Male or female adults ≥18 years of age.
2. Documented HIV-1 infection by Western Blot, Enzyme Immuno Assay (EIA) or viral load assay.
3. CMV seropositive (as per clinical lab test).
4. On ART for at least 3 years, and stable ART regimen (same prescription) for at least 3 months.
5. Undetectable viral load < 50 copies/ml for the past 3 years. Viral blips in the past 3 years, below 200 copies/ml, are allowed if preceded and followed by a HIV viremia below 50 copies/ml.
6. CD4 count >400 cells/µL of blood
7. Able to communicate adequately in either French or English.
8. Able to understand and willing to provide written informed consent prior to screening.
9. Women of childbearing potential must have a negative serum pregnancy test.
10. Women of childbearing potential must agree to use one of the following approved methods of birth control while in the study and until 2 weeks after completion of the study:

    Complete abstinence from penile-vaginal intercourse from the screening period until 2 weeks after study completion.

    Double barrier method (acceptable barrier methods include diaphragm, coil, contraceptive foam, sponge with spermicide, or condom).

    Oral, injectable or implant contraceptives, started at least 30 days before screening, plus one barrier method.

    Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion) plus one barrier method.

    Male partner sterilization confirmed prior to the female participant's entry into the study; this male is the sole partner for that participant.

    Another method approved by the Investigator with published data showing that the expected failure rate is <1% per year preferably with one barrier method.

    Any contraception method must be used consistently, in accordance with the approved product label, and for the duration of the study until two weeks after study completion.
11. Women of non-child-bearing potential as defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy.
12. Sexually active men with a female partner of childbearing potential must agree to one of the following methods of birth control:

The use of at least one barrier method of contraception (e.g. condom) with a female partner using a second approved method of contraception (IUD, hormonal contraceptive pill, diaphragm, spermicide, etc.) during the study and until two weeks after study completion.

Have had a successful vasectomy. Be confirmed sterile.

Exclusion Criteria:

Patients who are hypersensitive to letermovir or to any ingredient in the formulation of PREVYMIS®, including any non-medicinal ingredient, or component of the container.

Current AIDS-related event or serious health condition including systemic infections in the last 3 months.

Severe systemic diseases (e.g. uncontrolled hypertension, chronic renal failure), or active uncontrolled infections including Coronavirus disease 19 (COVID-19) (as tested by PCR).

Co-infection with active Hepatitis B or C Virus. Current use or have used in the past 3 months: immune-modulatory agents, prophylactic antibiotics, proton pump inhibitors, Metformin or Morphine as these drugs modulate inflammation and/or gut microbiota composition.

Current use of any drug with known drug-on-drug interaction with letermovir, as described in the PREVYMIS® (letermovir tablets) Product Monograph, including pimozide, ergot alkaloids, cyclosporine concomitantly administered with lovastatin, rosuvastatin, simvastatin or bosentan. For patients not using cyclosporine, dose of statins will be reduced by 50% for the duration of the study as a precaution, which is not expected to increase cardiovascular risk. Regarding HIV medication, exclusionary agents include darunavir, efavirenz, etravirine and nevirapine.

Recent changes in dietary habits, intermittent fasting, chronic constipation or laxative use as these can affect gut microbiota.

Psychiatric or cognitive disturbance or any illness that could preclude compliance with the study.

Current participation in an experimental therapy study or receipt of experimental therapy within the last 6 months.

Women who are planning to become or who are pregnant, or breast-feeding. A score of higher than 8 on a Full AUDIT questionnaire at the screening visit, suggesting an alcohol abuse problem.

Patients with moderate hepatic impairment combined with moderate or severe renal impairment (CrCl less than 50 mL/min)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Gut Inflammation | 28 weeks
  To assess the influence of CMV replication inhibition with letermovir on gut translocation markers (LPS) in blood of PLWH.

SECONDARY OUTCOMES:
Gut permeability | 28 weeks
  To assess the influence of CMV replication inhibition with letermovir on gut permeability markers in blood of PLWH (REG3α and I-FABP).
Inflammation markers | 28 weeks
  To assess the influence of CMV replication inhibition with letermovir on inflammation markers (IL-6, sCD14, hsCRP, d-dimers) in blood of PLWH.
Anti-CMV immune response | 28 weeks
  To assess the influence of CMV replication inhibition with letermovir o Anti-CMV immune response (anti-CMV IgG titers and specific T-cell response) and CMV DNA detection in plasma and PBMCs
CMV DNA detection in gut | 28 weeks
  To assess the influence of CMV replication inhibition with letermovir on in a sub-study, inflammation in colon biopsies obtained by coloscopy and in CMV DNA detection in gut mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Carolina A Berini, BSc, PhD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Mcgill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Royston L, Isnard S, Berini CA, Bu S, Lakatos PL, Bessissow T, Chomont N, Klein M, Lebouche B, de Pokomandy A, Kronfli N, Costiniuk CT, Thomas R, Tremblay C, Boivin G, Routy JP. Influence of letermovir treatment on gut inflammation in people living with HIV on antiretroviral therapy: protocol of the open-label controlled randomised CIAO study. BMJ Open. 2023 Jan 23;13(1):e067640. doi: 10.1136/bmjopen-2022-067640. PMID 36690406